CLINICAL TRIAL: NCT06578377
Title: The Epidemiology of Acute Respiratory Distress Among Children, A Retrospective Cross-Sectional Study From Iran
Brief Title: The Epidemiology of Acute Respiratory Distress Among Children, A Retrospective Cross-Sectional Study
Status: Completed | Type: Observational
Sponsor: Mofid Children Hospital (Other)
Collaborators: Dr Fatemeh Shojaeian, Dr seyed mohamadsadegh mousavi-kiasary, Dr Samira Sayyah (Unknown)
Responsible Party: Principal Investigator, Mahdis Bayat, Dr, Mofid Children Hospital
Other Study IDs: MofidCH
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Acute Respiratory Distress
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: descriptive study — It is a descriptive study

SUMMARY:
l Respiratory distress is still a major concern in pediatric medicine. l In this study we evaluated the symptoms and causes of respiratory distress among children in a tertiary hospital.

l We found that tachypnea is the most common symptom and asthma is the most common cause of respiratory distress in children.

ELIGIBILITY:
Inclusion Criteria:

* patients older than one month
* signs or symptoms of respiratory distress, including tachypnea, bradypnea, cyanosis, respiratory muscle retraction, nasal flaring, tachycardia, and bradycardia

Exclusion Criteria:

* Patients older than 18 years old
* apnea
* known cardiac diseases

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: From a total of 186 patients who visited the emergency room of Mofid Children's Hospital during the period of the study, 154 included in the study
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
The most common symptom | six months
The most common cause of respiratory distress | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Mahdis Bayat, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No